CLINICAL TRIAL: NCT01333735
Title: Impact on Cognitive Function and Quality of Life of Adjuvant Chemotherapy in Patients Aged Over 65 Years: Application to Breast Cancer or Colon
Acronym: COG AGE
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Collaborators: National Cancer Institute, France (Other Government); Sanofi (Industry)
Responsible Party: Pr Florence JOLY-LOBBEDEZ, Centre François Baclesse
Other Study IDs: COG AGE
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: cognitive functions; quality of life; breast cancer; chemotherapy; ages patients
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — NFS, uree, creatinin, ASAT, ALAT, PAL, GGT, Vit D, B12, Folates, Albumin, lipid, TSH, testosteron, oestradiol, LH, FSH, TP, TCA, D-Dimeres, Homocystéine, plasmatic biomarkers(protein S100, NSE, CRP, IL6)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with chemotherapy group: Patients with breast or colon cancer must beginning a chemotherapy (colon group was ended)
- Patients without chemotherapy group: patient with breast or colon cancer should not receive chemotherapy (colon group was ended)

SUMMARY:
The aim of the study is to investigate the impact of adjuvant chemotherapy on cognitive function in patients aged over 65 and suffering from breast cancer or colon.

ELIGIBILITY:
Inclusion Criteria for patients with chemotherapy :

* Patient(e) aged over 65 years
* Non metastatic breast cancer
* Adjuvant chemotherapy Breast cancer: FEC, including Docetaxel Protocols
* No major cognitive impairment
* Lack of personality disorders and psychiatric disorders evolutionary
* Having signed the informed consent of study participation

Inclusion Criteria for patients without chemotherapy (control group):

* Patient(e) aged over 65 years
* Breast cancer
* Patients receiving no adjuvant chemotherapy
* No major cognitive impairment
* Lack of personality disorders and psychiatric disorders evolutionary
* Having signed the informed consent of study participation
* Matching on age, sex, cultural level and tumor location

Exclusion Criteria for patients with chemotherapy :

* Metastatic
* Cancer primitive other than breast
* Patients under 65 years
* Patients with adjuvant chemotherapy is associated with targeted therapy
* Patients who have received other cancer treatments (chemotherapy or radiotherapy brain)
* disorders of higher functions existing in the administration of chemotherapy
* Pathology psychiatric evolutionary
* Refusal of participation
* Patients unable to meet the cognitive tests
* Drug use
* Heavy drinking

Min Age: 66 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients with chemotherapy group and patients without chemotherapy group (control group)
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2008-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
impact of memory impairment | Before chemotherapy (baseline), end of chemotherapy and follow-up up to 24 months after chemotherapy
  Assessing the impact of memory impairment induced by chemotherapy and study their evolution over time, with patients over 65 years treated in the adjuvant setting for breast cancer.
  Evaluated by auto-questionnary an tests with a neuropsychologist

SECONDARY OUTCOMES:
correlations between disorders of cognitive functions and parameters of quality of life | Before chemotherapy (baseline), end of chemotherapy and follow-up up to 24 months after chemotherapy
  Studying the correlations between disorders of cognitive functions and parameters of quality of life
Relationship between performance and onco-geriatric cognitive | Before chemotherapy (baseline), end of chemotherapy and follow-up up to 24 months after chemotherapy
  Examine the relationship between performance and onco-geriatric cognitive
Biological disturbances | Before chemotherapy (baseline), end of chemotherapy and follow-up up to 24 months after chemotherapy
  Search for biological disturbances may be related to cognitive impairment observed
Impact of age | Before chemotherapy (baseline), end of chemotherapy and follow-up up to 24 months after chemotherapy
  Assess the impact of age on the magnitude of cognitive impairment in patients
lived of the entourage | Before chemotherapy (baseline), end of chemotherapy and follow-up up to 12 months after chemotherapy
  - Assess the impact and cognitive impairment of patients'experiences of the circle (translational research)

CONTACTS AND LOCATIONS:
Overall Officials: Florence JOLY-LOBBEDEZ, PD, Principal Investigator — Centre François Baclesse
Locations (15):
- Université, Brussels, Belgium
- France (14):
  - INSERM, Caen, Calvados
  - CHU, Caen, Calvados
  - Centre François BACLESSE, Caen, Calvados
  - CHRU Hôpital Claude Huriez, Lille, Nord
  - Hopital gériatrique des Bateliers, Lille, Nord
  - Université, Lille, Nord
  - CHU, Hôpital Bois Guillaume, Rouen, Seine Maritime
  - CHU, Rouen, Seine Maritime
  - Centre Henri BECQUEREL, Rouen, Seine Maritime
  - Hôpital Charles FOIX, Ivry-sur-Seine
  - Hopitaux universitaires, Strasbourg
  - Hôpital Saint-Louis, Paris, Île-de-France Region
  - Hopital Pitié-Sapètrière, Paris, Île-de-France Region
  - Hopital TENON, Paris, Île-de-France Region